CLINICAL TRIAL: NCT03643432
Title: Can a Brief Behavioural Assessment Improve Exercise Adherence in Older People With Musculoskeletal Conditions: A Feasibility Randomised Controlled Trial
Brief Title: Adherence for Exercise Rehabilitation in Older People Trial
Acronym: AERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Jonathan Room, Senior Research Physiontherapist, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13594
Record Dates: First submitted 2018-05-22; First posted 2018-08-22 (Actual); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Geriatric; Exercise Adherence

STUDY DESIGN:
Intervention Model Description: Participants will be randomised between usual care or the intervention arm which will consist of a brief behavioural assessment and recommended adherence strategies based on the outcome of the assessment. A sub sample of the population will undergo a qualitative study to assess acceptability of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): The usual care arm will consist of routine physiotherapy treatment, without the intervention.
  Interventions: Behavioral: Usual Care
- Exercise adherence intervention (Experimental): The intervention arm will consist of a brief behavioural assessment and recommended adherence strategies based on the outcome of the assessment.
  Interventions: Behavioral: Exercise adherence intervention

INTERVENTIONS:
Behavioral: Exercise adherence intervention — Before their physiotherapy appointment participants will be given four short questions to answer. Following this the participant will be assessed as normal. As part of the treatment they will be given an exercise programme as standard within physiotherapy. Following this participants will be asked to answer a further seven short questions; depending on the answers to both sets of questions, and on any discussion based on the answers, the physiotherapist will suggest one or more adherence approaches from a list of suggestions. These are; Review of exercise programme; Review of method of delivery; Cues or prompts; Discussion of barriers and problem solving; Motivational interviewing, Decision balance sheets; Behavioural contract; Goal setting review; Monitoring telephone call; Reminders.
  Arms: Exercise adherence intervention
Behavioral: Usual Care — Participants in usual care will attend physiotherapy sessions as they would have had they not been in the trial.These sessions will include assessment and treatment approaches as given as part of routine care, without including the intervention described above for the 'exercise adherence intervention' arm
  Arms: Usual care

SUMMARY:
Exercise is an effective treatment modality for many chronic conditions. The effectiveness of prescribed exercise can be limited by adherence to exercise programmes. Older people are more likely to have a long term, or multiple long term conditions, for which exercise is a treatment option. The investigators know that exercise engagement after discharge from hospital or physiotherapy is poor in older people. In addition to this there may be specific factors that affect exercise adherence in older people. Exercise adherence interventions can be viewed as behaviour change interventions, as their aim is to change the behaviour of the patient. However many interventions lack theoretical underpinning. This study will test the feasibility of a brief behavioural assessment underpinned by the COM-B behaviour change model, in addition to targeted adherence approaches based on that assessment. Participants will be randomised between usual care, and the behavioural assessment intervention arm. Adherence to the exercise programme given in physiotherapy will be recorded in both groups at 6 and 12 weeks. Feasibility of recruitment, retention and acceptability of the intervention will also be assessed. A subsection of participants will also take part in a qualitative interview, this will explore participants experience of the trial intervention, in addition to the participants experience of attempting to adhere to an exercise programme.

DETAILED DESCRIPTION:
The design of this study, is a a two arm feasibility randomised controlled trial. Participants will be randomised between usual care, or the intervention arm which will consist of a brief behavioural assessment and recommended adherence strategies based on the outcome of the assessment. A sub sample of the population will undergo a qualitative interview to assess acceptability of the intervention

Potential research participants will be invited to take part in the study with an invitation letter, along with the PIS and a reply slip. These will be sent out with information about their physiotherapy appointment, which they would normally receive.

After time to consider the study and ask any questions, if participants are happy to take part, an appointment will be made to take consent and collect baseline measures. This will take place at the Nuffield Orthopaedic Centre, if possible just prior to their physiotherapy appointment in order to limit disturbance to the participant. If this is not possible the appointment to collect consent and baseline data will be at a time convenient to the patient. At this appointment, signed consent will be recorded and baseline data collected. This will involve the participants completing some questionnaires.

Treatment allocation will be decided on the basis of the physiotherapist the participant is seeing. (Before the start of the study all physiotherapist taking part in the study will be randomly assigned to deliver either usual care or the intervention arm). Those participants in usual care will undergo physiotherapy as normal, the only additional thing they will be asked to do, is to complete an exercise diary for up to 12 weeks.

Those in the intervention arm will be asked to complete 4 short questions related to exercise and treatment expectations. These will be completed in the waiting room prior to the physiotherapy appointment. The participant will be assessed and given treatment as normal in physiotherapy. After they have been given an exercise programme as part of their treatment, they will be asked to complete a further 7 short questions related to the exercise programme, and their motivation and intention to undertake it. On the basis of the answers to these questions and also in addition to any discussion with the physiotherapists, one or more adherence approaches may be suggested. The approaches are 'review of exercise programme', 'review of method of delivery', 'cues', 'reminders', 'discussion of barriers and problem solving', 'motivational interviewing', 'decision balance sheets', 'behavioural contract' and 'goal setting review'. The participants in the intervention group will also be asked to complete an exercise diary for up to 12 weeks.

Participants in both groups will be followed up at 6 weeks and 12 weeks after their initial physiotherapy appointment. the follow appointment will consist of completing some questionnaires and to collect exercise diaries (12 week follow up). For the majority of participants this will be the end of the study. However a small sub-sample of participant will be invited to take part in an interview. This will last no longer than 1 hour, and will aim to explore the views of participants regarding the study, and also about trying to stick to an exercise programme. Participants will be given time to consider taking part in this additional interview, and will be asked to provide signed consent. Once they have finished the interview, they will be finished in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 65 years or above
* Referred to physiotherapy with a musculoskeletal problem
* Able to converse in and read English

Exclusion Criteria:

* Any comorbidity that precludes exercising such as unstable angina, or acute illness
* Dementia or cognitive impairment precluding the ability to follow an exercise programme
* Patients referred to physiotherapy for post-surgery rehabilitation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan F Room, MRes, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Nuffield Orthopaedic Centre, Oxford University Hospitals NHS FT, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Room J, Dawes H, Boulton M, Barker K. The AERO study: A feasibility randomised controlled trial of individually tailored exercise adherence strategies based on a brief behavioural assessment for older people with musculoskeletal conditions. Physiotherapy. 2023 Mar;118:88-96. doi: 10.1016/j.physio.2022.08.006. Epub 2022 Aug 30. PMID 36266133

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Exercise Adherence Intervention
Started | 27 | 21
Completed | 26 | 21
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Exercise Adherence Intervention | Total
Number analyzed (Participants) | 26 | 21 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 26 | 21 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.58 (7.05) | 74.10 (6.20) | 74.36 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 26 | 21 | 47
Tilburg Frailty Indicator [Mean (Standard Deviation); unit: units on a scale] — Tilburg Frailty Index. Scale, with a possible score ranging from 0 to 15 with a higher score being more indicative of frailty, a cut point of 5 is suggested in order to consider an individual as frail.
  units on a scale | 5.04 (3.34) | 4.86 (3.41) | 4.96 (2.84)
Physical Activity Scale for the Elderly (PASE) [Mean (Standard Deviation); unit: units on a scale] — The range of the score depends on the amount of work that a participant does, a higher score indicates an individual who is more physically active
  units on a scale | 137.61 (82.67) | 112.50 (70.08) | 126.38 (82.67)
Self-efficacy for exercise scale [Mean (Standard Deviation); unit: units on a scale] — This scale measures self-efficacy expectations to continue to exercise in the face of barriers to exercise. Scores can range from 0-90, with higher scores indicating greater self-efficacy for exercise.
  units on a scale | 64.69 (21.52) | 59.14 (19.43) | 62.21 (20.58)
Self-rated capacity to exercise [Mean (Standard Deviation); unit: units on a scale] — Self-rated capacity to exercise was scored on a Visual Analogue Scale (VAS), participants were asked to rate their perceived capacity to exercise on a scale of 0-10, where 0 is no capacity and 10 is maximum capacity
  units on a scale | 6.77 (2.47) | 6.48 (2.66) | 6.64 (2.53)
Self-rated confidence to exercise [Mean (Standard Deviation); unit: units on a scale] — Self-rated confidence to exercise was scored on a Visual Analogue Scale (VAS), participants were asked to rate their perceived confidence to exercise on a scale of 0-10, where 0 is no confidence and 10 is maximum confidence.
  units on a scale | 7.35 (2.56) | 6.48 (2.58) | 6.96 (2.58)
Self-rated motivation to exercise [Mean (Standard Deviation); unit: units on a scale] — Self-rated motivation to exercise was scored on a Visual Analogue Scale (VAS). Participants were asked to rate their perceived motivation to exercise on a scale of 0-10, where 0 is no motivation and 10 is maximum motivation.
  units on a scale | 7.85 (2.54) | 7.29 (2.43) | 7.60 (2.48)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Adherence
Description: This is a self-report scale ranging from 0-10, where patient will be asked to rate their adherence over the previous twelve weeks, ranging from 0 = 'no exercises performed' to 10 = 'all exercise performed as instructed'
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 26 | 21
score on a scale
  6 weeks | 6.77 (2.86) | 7.35 (3.00)
  12 weeks | 6.60 (3.00) | 7.10 (2.77)

2. Secondary Outcome: Exercise Adherence Rating Scale (EARS)
Description: The Exercise Adherence Rating Scale is a 6 item self-report questionnaire, that asks people to record the answer to 6 question on exercise adherence, on a 5 point Likert scale. Each question is scored 0 to 4 (0 - completely agree to 4 - completely disagree), however questions 1,4 and 6 are reverse scored (4 - completely agree to 0 - completely disagree). The total score can range from 0-24. A higher score equals better adherence.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 26 | 21
score on a scale
  6 weeks | 16.35 (5.87) | 18.25 (5.82)
  12 weeks | 15.64 (6.60) | 17.38 (6.78)

3. Secondary Outcome: Exercise Diary
Description: This diary will have been completed post physiotherapy, recording the number, sets and reps of exercises that the patient has been undertaken.
Time Frame: 12 weeks
Population: Some participants lost their diaries and did not return them at follow up, therefore 21 in usual care were analysis and 16 in the intervention arm were analysed.
Measure: Mean (Standard Deviation); unit: percentage of completed exercise
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 21 | 16
percentage of completed exercise | 62.57 (27.47) | 77.21 (18.33)

4. Secondary Outcome: Global Rating of Change
Description: This is the participants' perception of their change since their initial appointment; possible scores range from -3 = 'very much worse', -2 = 'much worse', -1 = 'a little worse', 0 = 'about the same/no difference', 1 = 'a little better', 2 = 'much better', 3 = 'very much better'. Higher scores indicate a better outcome.
Time Frame: 6 weeks and 12 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 26 | 21
units on a scale
  6 weeks | 1 [-3 to 3] | 1 [-3 to 3]
  12 weeks | 1 [-3 to 3] | 1 [-3 to 3]

5. Secondary Outcome: Physical Activity Scale for the Elderly (PASE)
Description: The Physical Activity Scale for the Elderly is a physical activity self-report questionnaire that takes around 5-10 minutes to complete. Different activities have been weighted as assigned by the developers of the scale. The total score for PASE is calculated by multiplying the time spent undertaking an activity by it's respective weigh. Scores range from 0 to 360, with higher scores equating to more physical activity.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 26 | 21
score on a scale
  6 weeks | 132.96 (70.75) | 131.48 (70.68)
  12 weeks | 132.45 (70.86) | 137.14 (98.57)

6. Secondary Outcome: EQ 5D 5L
Description: This self-report questionnaire is a measure of health-related quality of life. Scores for each question range from 1 to 5, these scores are converted to an index value ranging from -0.5940 to 1.0000, a higher score indicating a better health state
Time Frame: 6 weeks and 12 weeks
Population: Numbers analysed different at 6 and 12 weeks due to sections of questionnaires not completed by 2 participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 26 | 21
units on a scale
  6 weeks: number analyzed (Participants) | 26 | 19
  6 weeks | 0.632308 (0.1499250) | 0.618553 (0.2104626)
  12 weeks | 0.645892 (0.1544202) | 0.600624 (0.3110265)

7. Secondary Outcome: Self-Efficacy for Exercise Scale
Description: The Self-Efficacy for Exercise Scale is a self-report scale that measures self-efficacy expectations to continue to exercise in the face of barriers to exercise. It consists of 9 questions each scored from 0 to 10, this gives a total score range of 0 to 90. A higher score indicates higher self-efficacy for exercise.
Time Frame: 6 weeks and 12 weeks
Population: At 12 weeks, 2 questionnaires had SEE left blank
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 26 | 21
score on a scale
  6 weeks | 61.50 (22.83) | 61.00 (22.07)
  12 weeks: number analyzed (Participants) | 26 | 19
  12 weeks | 58.20 (23.58) | 52.53 (28.16)

8. Secondary Outcome: Exercise Regulations Questionnaire (BREQ-3)
Description: This self-report questionnaire measures motivation for exercise, it measures forms of intrinsic and extrinsic regulation of exercise behaviour. It consists of 24 questions, each question is scored from 0 to 4, these scores can be summed to give various subscale scores, or all questions can be used by summing scores and multiplying by its subscores weighing to obtain the relative autonomy index (RAI) score. The RAI score can range from -24 to 24. A higher score indicating greater relative autonomy and a lower score indicating more controlled regulation.
  higher scores indicates more relative automony, and lower scores a more controlled regulation.
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 26 | 21
units on a scale
  6 weeks | 9.27 (8.36) | 11.55 (8.25)
  12 weeks | 8.56 (9.40) | 9.71 (8.31)

9. Secondary Outcome: VAS Self-rated Capacity to Exercise, Confidence to Exercise and Motivation to Exercise
Description: Participants will be asked to rate their perceived capacity, confidence and motivation to exercise on a scale of 0-10, where 0 is no capacity/confidence/motivation' and 10 is maximum capacity/confidence/motivation
Time Frame: 6 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Exercise Adherence Intervention
Number analyzed (Participants) | 26 | 21
score on a scale
  6 weeks Capacity | 7.85 (2.05) | 7.00 (2.73)
  12 weeks Capacity | 7.44 (2.60) | 7.48 (2.48)
  6 weeks Confidence | 8.00 (2.26) | 7.50 (2.95)
  12 weeks confidence | 7.48 (2.84) | 7.48 (2.84)
  6 weeks Motivation | 8.15 (2.13) | 8.05 (2.54)
  12 weeks Motivation | 8.00 (2.31) | 7.57 (2.82)

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Arm/Group | Usual Care | Exercise Adherence Intervention
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/21
Other Adverse Events (participants affected / at risk) | 0/26 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT03643432/Prot_SAP_000.pdf